CLINICAL TRIAL: NCT06638463
Title: Randomized Controlled Trial of the My Health Coach App for Adults With Fetal Alcohol
Brief Title: My Health Coach App RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Christie Petrenko, Director of Clinical Training, Department of Psychology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00009709
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Fetal Alcohol Spectrum Disorders
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- My Health Coach App Group (Experimental): The My Health Coach group receives the My Health Coach app at study start. The My Health Coach app is a self-directed mobile health intervention for adults with FASD. It is grounded in self-determination theory and integrates well-established behavior change strategies. It has a cloud-based infrastructure and uses a just-in-time adaptive intervention design and a simple and engaging chatbot interface. It provides adults just the right type and amount of support, when they are most receptive.
  Interventions: Behavioral: My Health Coach app
- Waitlist Control Group (No Intervention): The Waitlist Control Group gets access to the My Health Coach app after all the study survey timepoints are complete at 12 weeks.

INTERVENTIONS:
Behavioral: My Health Coach app — My Health Coach is a self-directed mobile health intervention for adults with FASD. It is grounded in self-determination theory and integrates well-established behavior change strategies. It has a cloud-based infrastructure and uses a just-in-time adaptive intervention design and a simple and engaging chatbot interface. It provides adults just the right type and amount of support, when they are most receptive.
  Arms: My Health Coach App Group

SUMMARY:
The goal of this clinical trial is to learn if the My Health Coach app helps adults with fetal alcohol spectrum disorders (FASD). The main questions it aims to answer are:

Does the My Health Coach app improve the quality of life of adults with FASD? Does the My Health Coach app help adults with FASD manage their day to day life?

All participants will be asked to complete 3 sets of surveys: 1) at the study start, 2) at 6 weeks, and 3) at 12 weeks. Half of the participants will be given the app at the study start to use. The other half of participants will get the app after the 12 week surveys are complete.

Researchers will compare survey results from people who receive the app right away to those who are in the waitlist group to see if there are changes in quality of life or day to day functioning.

DETAILED DESCRIPTION:
This trial involves a 2-arm randomized controlled trial. Participants will be randomized (50:50 allocation) into the (1) My Health Coach group, or the (2) Wait-list Control group. The My Health Coach app is designed to support the quality of life of adults with FASD by providing tools to help with self-management, advocacy, health literacy, use of supports, and engagement in meaningful activities.

This study is designed to: (1) evaluate the efficacy of the My Health Coach app with adults with FASD, (2) test whether changes in competence, autonomy, and/or relatedness mediate intervention outcomes on reported quality of life, and (3) identify app usage patterns that relate to greater outcome improvement. Primary outcomes include perceived well-being, the degree to which basic psychological needs of competence, autonomy, and relatedness are met, and readiness for self-management. We are also interested in participants' perceptions of app quality and patterns of app usage.

All participants will complete the study assessment battery measuring these outcomes at baseline (T1), 6 weeks (T2), and 12 weeks (T3). Wait-list participants will receive the app after T3.

ELIGIBILITY:
Inclusion Criteria:

* adult 18 years or older
* have a fetal alcohol spectrum disorder (FASD) or history of prenatal alcohol exposure
* have sufficient fluency in written English
* own a smartphone

Exclusion Criteria:

* participated in the past feasibility trial of the My Health Coach app

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean effect size on the Personal Well-being Index - Intellectual Disability Version (complemented by statistical hypothesis testing and 95% CI) | Baseline to 12 weeks
  The PWI is an 8-item measure of subjective wellbeing. The Intellectual Disability Version uses more concrete item wording and a 5-point pictoral scale. Ratings are summed and higher scores reflect better perceived well-being. An effect size of 0.2 is small, 0.5 is medium, and 0.8 is large.
Mean effect size on The Basic Psychological Need Satisfaction and Frustration Scale (complemented by statistical hypothesis testing and 95% CI) | Baseline to 12 weeks
  The BPNSF is a 24-item scale assessing both satisfaction and frustration relating to the three basic psychological needs identified in self-determination theory: autonomy, competence, and relatedness. Items are rated on a 5-point scale from 1 "not at all true" to 5 "completely true." Higher scores reflect higher satisfaction or need being met to a higher degree. An effect size of 0.2 is small, 0.5 is medium, and 0.8 is large.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes